CLINICAL TRIAL: NCT04994353
Title: Pre-meal High-performance Inulin Supplementation Reduce Post-prandial Glycaemic Response in Healthy Non Diabetic Subjects : a Repeated Single-arm Clinical Trial
Brief Title: Pre-meal High-performance Inulin Supplementation in Healthy Non-diabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Katolik Widya Mandala Surabaya (Other)
Responsible Party: Principal Investigator, Hendy Wijaya, MD, Universitas Katolik Widya Mandala Surabaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 131/WM12/KEPK/DOSEN/T/2020
Record Dates: First submitted 2021-07-27; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Diet, Healthy
Keywords: high performance inulin; glycaemic index; blood glucose; pre-meal; post-prandial
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supplementation (Experimental): Three days before the intervention, every subject was informed to maintain their normal diet, physical activities, and enough sleep (6-8 hours/day). All subjects fasted 10-12 hours before the intervention. An intravenous cannula was inserted into the cubital vein to provide access to repeated glucose measurement. Peripheral vein whole blood samples were taken for analysis of glucose concentration using a commercially available FreeStyle Optium glucose monitoring system (Abbot Laboratories, Chicago, Illinois, USA) .For the first week, we measured blood glucose to a meal without any intervention and use those data as a baseline. After that, blood glucose was measured at 0, 30, 60, 90, and 120 minutes after intervention and meal. After intervention, the subjects maintain daily predefined ready-meal (470 kcal). The supplementation formulas are "food grade", purchased from PT. Lautan Natural Krimerindo (Mojokerto, Jawa Timur, Indonesia).
  Interventions: Dietary Supplement: No supplementation; Dietary Supplement: High Performance (HP) Inulin; Dietary Supplement: Isomalto-oligosaccharide (IMO); Dietary Supplement: Combination HP-Inulin and IMO; Dietary Supplement: Dextrose solution; Dietary Supplement: Glucose solution

INTERVENTIONS:
Dietary Supplement: No supplementation — 1st Week: No supplementation
Dietary Supplement: High Performance (HP) Inulin — 2nd Week: Subjects consumed 20% v/v HP Inulin. Ingredients: 20 gram HP-Inulin diluted with 100 ml distilled water.
Dietary Supplement: Isomalto-oligosaccharide (IMO) — 3rd Week: Subjects consumed 20% v/v Isomalto-oligosaccharide (IMO). Ingredients: 20 gram IMO diluted with 100 ml distilled water.
Dietary Supplement: Combination HP-Inulin and IMO — 4th Week: Subjects consumed20% v/v combination of HP-Inulin and Isomalto-oligosaccharide (IMO).
  Ingredients: 20 gram IMO-HP Inulin "Mix" diluted with 100 ml distilled water.
Dietary Supplement: Dextrose solution — 5th Week:Subjects consumed20% v/v Dextrose solution. Ingredients: 20 gram Dextrose powder diluted with 100 ml distilled water.
Dietary Supplement: Glucose solution — 6th Week:Subjects consumed 20% v/v Glucose solution. Ingredients: 20 gram glucose diluted with 100 ml distilled water.

SUMMARY:
In a double-blind, repeated single-arm trial, 8 healthy adults consumed 20 grams of formula that contain 60.2% inulin (w/w) dissolved in 100 ml of water. Blood glucose was measured in fasted participants and at, 30, 60, 90, and 120 minutes after starting to eat a prepared meal (470 Kcal). As supplementation controls, the investigators used the vehicle-glucose, dextrose, isomaltooligosaccharides (IMO), or the combination of IMO and Inulin solution 20% (w/v).

DETAILED DESCRIPTION:
Subjects In this trial, 8 healthy subjects (6 women and 2 men), aged between 23-37 years old were voluntarily recruited. Inclusion criteria were: healthy men or women aged between 18-50 years old, body mass index (BMI) between 18.5-25.0, normal diet, not under any medication, and not having any history of metabolic diseases or abnormalities such as systemic hypertension (resting blood pressure more than 140/90 mmHg), impaired glucose tolerance (fasting blood glucose concentration between 100-126 mg/dL and oral glucose tolerance test or OGTT more than 140 mg/dL), and non-alcoholic fatty liver diseases (NAFLD). Subjects were excluded if they had an acute infection, pregnant, gastrointestinal disease, cardiovascular disease, renal disease, pancreatic disease, and take any medication during or 1 week before trial. At the beginning of the trial, demographic data including age, sex, history of diseases, medication, diet, and physical activities within 3 days were collected using a questionnaire form. Bodyweight was measured using Omron digital scale HN286 (PT. Omron Manufacturing of Indonesia). Body height was measured using a stature meter. To determine the amount of daily calorie expenditure for selection of the suitable ready-meal, the estimated energy requirements (EER) were calculated based on the harris-benedict formula as previously reported45, with the physical activity level 1.0 (sedentary activity). This research was approved by the Health Research Ethics Committee of Widya Mandala Catholic University Surabaya (No. 131/WM12/KEPK/DOSEN/T/2020).

Experimental design This experimental design adapted a single-arm trial analysis. A group of 8 subjects received intervention with single pre-meal supplementation. After that, the glycaemic response was measured (see blood sampling preparation). This intervention was repeated every week with five different supplementation formulae (see below) for five consecutive weeks. The difference in their glycaemic response after meal for every intervention was measured and analyzed statistically.

Supplement preparation: Inulin formulations, isomaltooligosaccharides formulations, the combination of inulin and isomaltooligosaccharides formulations, dextrose solution, and vehicle-glucose formulations.

For the first week, the investigators measured glycaemic response to a meal without any intervention and use those data as a baseline. For the intervention, the investigators used the untreated control without supplementation (NS), HP Inulin formulations (IF), isomaltooligosaccharides/IMO formulations (IM, this formulation is marketed as Fibercreme®), the combination of HP inulin and IMO formula (MF), dextrose solution (DS), and vehicle-glucose formulations (VO) in the form of powder. All the supplementation formulas are purchased from PT. Lautan Natural Krimerindo (Mojokerto, Jawa Timur, Indonesia). The detailed composition of each formulation could be seen in Supplementary Table 1. For the preparation of 20% IF, IM, and MF solution, 20 grams of designated powder was diluted in 100 ml distilled water. For 20% DS, 20 grams of purified dextrose monohydrate was diluted in 100 ml distilled water. IMO solution was chosen as a control because IMO could act as partially digestible dietary fibre.43 Vehicle-glucose could act as a negative control for IF intervention because IF contains similar ingredients with the IF, but instead of inulin, glucose syrup was added as the caloric source.

Intervention: fasting, pre-meal supplementation, and meal Three days before the intervention, every subject was informed to maintain their normal diet, physical activities, and enough sleep (6-8 hours/day). All subjects fasted 10-12 hours before the intervention. Supplement formula solution 20% (w/v) then given orally before a meal for five consecutive weeks in the following orders: IF in the first week, followed by IM in the second week, MF in the third week, DS in the fourth week, and VO in the last week. The meal for experimental subjects was given after intervention and contained 470 kcal "Ready Meal". The amount of calories in "Ready-Meal" is 25-30% from the calculated EER (see table 1). The macronutrient composition of the "Ready Meal" was purchased from PT. Charoen Pokphand Indonesia,TbK (Jakarta, Indonesia) was listed in supplementary table 2.

Blood sampling preparation, blood glucose, and glycaemic response (iAUC) measurement.

An intravenous cannula was inserted into the cubital vein to provide access to repeated glucose measurement. Peripheral vein whole blood samples were taken for analysis of glucose concentration using a commercially available FreeStyle Optium glucose monitoring system (Abbot Laboratories, Chicago, Illinois, USA). Blood glucose was measured at 0, 30, 60, 90, and 120 minutes after intervention and meal. The first measurement at 0 representing the fasting plasma glucose (FPG), that is the blood glucose concentration after an overnight fast (10-12 hours). The glycaemic response measurement unit at 0, 30, 60, 90, and 120 minutes for each subject was described as the incremental area under the curve (iAUC). The iAUC refers to actual body exposure to certain substances after their administration. The AUC depends on the rate of substance elimination from the body and its dose of administration. iAUC calculation (symbolized with A) was carried out using a linear trapezoidal method and formula (see supplementary figure 1) as described in the literature.44

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 18.5-25.0
* normal diet
* not under any medication
* not having any history of metabolic diseases
* not having abnormalities such as systemic hypertension (resting blood pressure more than 140/90 mmHg), impaired glucose tolerance (fasting blood glucose concentration between 100-126 mg/dL and oral glucose tolerance test or OGTT more than 140 mg/dL), and non-alcoholic fatty liver diseases (NAFLD).

Exclusion Criteria:

- Subjects were excluded if they had an acute infection pregnant, gastrointestinal disease, cardiovascular disease, renal disease, pancreatic disease, and take any medication during or 1 week before trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Blood Glucose at T=0 | 0 minutes after intervention and meal
  Postprandial Blood glucose concentration
Blood Glucose at T=30 min | 30 minutes after intervention and meal
  Postprandial Blood glucose concentration
Blood Glucose at T=60 min | 60 minutes after intervention and meal
  Postprandial Blood glucose concentration
Blood Glucose at T=90 min | 90 minutes after intervention and meal
  Postprandial Blood glucose concentration
Blood Glucose at T=120 min | 120 minutes after intervention and meal
  Postprandial Blood glucose concentration

CONTACTS AND LOCATIONS:
Overall Officials: Hendy Wijaya, MD.M.Biomed., Principal Investigator — Faculty of Pharmacy, Universitas Katolik Widya Mandala Surabaya
Locations (1):
- Universitas Katolik Widya Mandala Surabaya, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murray CJ, Vos T, Lozano R, Naghavi M, Flaxman AD, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gonzalez-Medina D, Gosselin R, Grainger R, Grant B, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Laden F, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Levinson D, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mock C, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiebe N, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, AlMazroa MA, Memish ZA. Disability-adjusted life years (DALYs) for 291 diseases and injuries in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2197-223. doi: 10.1016/S0140-6736(12)61689-4. PMID 23245608
- [Background] GBD 2016 Causes of Death Collaborators. Global, regional, and national age-sex specific mortality for 264 causes of death, 1980-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1151-1210. doi: 10.1016/S0140-6736(17)32152-9. PMID 28919116
- [Result] Lambadiari V, Korakas E, Tsimihodimos V. The Impact of Dietary Glycemic Index and Glycemic Load on Postprandial Lipid Kinetics, Dyslipidemia and Cardiovascular Risk. Nutrients. 2020 Jul 24;12(8):2204. doi: 10.3390/nu12082204. PMID 32722053